CLINICAL TRIAL: NCT02440945
Title: Use of the DBS for the Follow-up of Blood Clinical Parameters of Old People
Acronym: DBSage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9114
Record Dates: First submitted 2015-04-16; First posted 2015-05-12 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- collection of blood (Experimental): 160 old people for the collection of blood
  Interventions: Device: Collection of blood

INTERVENTIONS:
Device: Collection of blood — Blood test on blotting paper DBS (for the patients recruting)

SUMMARY:
It is about an interventional study.The use of the blotting paper called "Dried Blood Spot" or DBS is a method of systematic neonatal screening of the metabolic diseases. Indeed, it has multiple interests: realized thanks to lancets, it is much less invasive than a classic blood collection. Besides, the transport of the blood sampling is facilitated because most of the analysts are stable on DBS at room temperature one week or more. Finally the use of this DM reduces the infectious risks bound to the manipulation of the blood sampling and to the inactivation of microorganisms. The moderate results are vitamin D, albumin, prealbumin, CRP, orosomucoide

The DBS presents a major interest for the care of the old and fragile people who have on one hand a low peripheral venous capital and on the other hand for whom the possibility of a dosage on DBS will allow a facilitated biological follow-up. Indeed it is very important to detect as soon as possible the most fragile old people, those who have the biggest risk of seeing their health degrading during a physical, psychic or social stress, to concentrate the efforts of coverage and limit these risks. The advantage of the biological criteria is the speed of the test making (a blood test), in the absence of necessity of active participation by the patient (the clinical criteria require to test the patient in the walking, to test its muscular strength, etc.) and in the saving of time diagnosis for the clinician. The blood biological markers of the fragility are essentially the rate of 25OH vitamin D, the markers of undernutrition (albumin, prealbumin) and of the inflammation (CRP, orosomucoïde). These last four parameters are now measurable from the DBS thanks to the quantitative mass spectrometry.

DETAILED DESCRIPTION:
Main objective: Define the analytical concordance between dosages realized on blotting paper (DBS) and classic dosages after blood test for the five markers.

Secondary objectives: Study the influence of the hématocrite, the hemoglobin, the total proteins on the dosages on DBS, and realize a biological collection of blood sample on DBS.

Methods and Feasibility:

The recruitment of the patients will be made with the Service of Geriatrics of the CHRU of Montpellier (Pr C. Jeandel, Dr G. Baptista), which have an important number of compatible patients with the number of planned patients for the study. In the standard blood results will be added a capillary taken which will be deposited on 3 DBS. The study of concordance of biological methods will include on one hand an analytical evaluation of the new methods in terms of reproducibility, repeatability, limit of detection and quantification. On the other hand, a comparison of the values of the dosages on venous taking (blood test) for normal and pathological values will be realized by the method of Bland and Altman associated with a regression of balanced Deming.

Calendar of the study:

M0-M6: optimization of the analytical method / M0-M3: Statutory for the clinical part (CPP..) M4-M16: inclusion of the patients / M6-M20: validation of the dosages on DBS M12-M24: valuation of the results (scientific articles, presentations, exploit the know-how)

Perspectives :

To be able to realize thanks to the DBS the follow-up of these biological parameters at the old people is a major step forward for the patients by avoiding classic blood test and by facilitating the preanalytical phase, making it more easily compatible with the telemedicine in particular, with the dosages practicable at home, in retirement home, at the doctor's office, with simple postal sending to analysis laboratories.

ELIGIBILITY:
inclusion criteria:

* Man / woman
* Having a standard blood test planned during their consultation or their hospitalization in the service of Geriatrics of Pr C. Jeandel
* Signature of the informed consent by the patient
* Patient affiliated to a national health insurance exclusion criteria:
* Absence of signed informed consent
* Patients with cutaneous disorders which increase the risks caused by the blood test (cutaneous infection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2015-10-16 (Actual); Study Completion 2015-10-16 (Actual)

PRIMARY OUTCOMES:
Use of the DBS for the follow-up of blood clinical parameters of the old people | 36 months
  The moderate results are vitamin D, albumin, Prealbumin, CRP, Prealbumin, orosomucoide CRP, Orosomucoide

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain lehmann, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHRU, Montpellier, France

REFERENCES:
- [Background] Tall ML, Lehmann S, Diouf E, Gerard C, Filali S, Gabelle A, Hirtz C, Gabert L, Sauvinet V, Pirot F, Pivot C. [Injectable preparation of labeled leucine with the carbon 13 for a clinical research program on the Alzheimer disease: pharmaceutical control of raw materials and the finished product and stability study]. Ann Pharm Fr. 2015 Jan;73(1):43-59. doi: 10.1016/j.pharma.2014.06.002. Epub 2014 Jul 11. French. PMID 25577016